CLINICAL TRIAL: NCT00687063
Title: An Observational, Safety and Efficacy Study in Subjects Using Levemir® (Insulin Detemir) for the Treatment of Type 2 Diabetes Mellitus.
Brief Title: Observational Study of Safety and Efficacy of Levemir® in Type 2 Diabetes
Acronym: DIABESITY
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3530
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency of insulin detemir is to be decided by physician. The choice of patient is also at the discretion of Physician
  Other Names: Levemir®

SUMMARY:
The study is conducted in Asia. The aim of this observational study is to evaluate the weight change from baseline while using Levemir® in subjects with type 2 diabetes mellitus under normal clinical practice conditions in India.

ELIGIBILITY:
Inclusion Criteria:

* Any subject with type 2 diabetes

Exclusion Criteria:

* Subjects with a hypersensitivity to insulin detemir or any of its excipient
* Children below 6 years
* Subjects who are pregnant, lactating or planning to become pregnant

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetics
Sampling Method: Non-Probability Sample
Enrollment: 10008 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Weight change from baseline | after 26 weeks

SECONDARY OUTCOMES:
Number of serious adverse events | after 26 weeks
Number of all adverse events | after 26 weeks
Number of all hypoglycemic episodes (24 hr, daytime and nocturnal) | after 26 weeks
HbA1c change from baseline | after 26 weeks
FBG (Fasting Blood Glucose) change from baseline | after 26 weeks
Percentage of patients achieving targets of HbA1c less than 7 % and less than 6.5 % | after 26 weeks
Insulin dose and frequency at the end of the study | after 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), MD, Study Director — Novo Nordisk A/S
Locations (1):
- Bangalore, India

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com